CLINICAL TRIAL: NCT03427944
Title: the Effect of Calcium Dobesilate on Non Dialysis Patients With Chronic Renal Failure
Brief Title: the Effect of Calcium Dobesilate on Non Dialysis Patients With CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL001-02
Record Dates: First submitted 2018-01-17; First posted 2018-02-09 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Chronic Renal Failure
Keywords: Calcium Dobesilate; Non Dialysis Patients With CKD(3-5); Glomerular filtration rate; serum creatinine
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium Dobesilate group (Active Comparator): Calcium dobesilate group was treated with calcium dobesilate (500mg, tid , po), its conservative treatment was the same as that of the conventional treatment group
  Interventions: Drug: Calcium Dobesilate group
- Conventional Treatment group (Placebo Comparator): conventional treatment group was treated with conventional conservative treatment of renal failure (low protein, low salt, low fat, low phosphorus diet, balance the internal environment; control blood pressure ; remove intestinal toxins etc.)
  Interventions: Drug: Conventional Treatment group

INTERVENTIONS:
Drug: Calcium Dobesilate group — Calcium dobesilate was used to treat patients with chronic renal failure on the basis of conventional treatment.
  Other Names: Treatment group
  Arms: Calcium Dobesilate group
Drug: Conventional Treatment group — Conventional treatment were used to treat patients with chronic renal failure.
  Other Names: Control group
  Arms: Conventional Treatment group

SUMMARY:
To investigate the feasibility of calcium dobesilate in the treatment of microvascular injury provides new ideas and theoretical basis for the prevention and treatment of chronic renal failure.

DETAILED DESCRIPTION:
The deterioration of renal function is closely related to microvascular damage, calcium dobesilate is known as microcirculation protective agent, the investigators will further study its effect of non dialysis patients with chronic renal failure and explore the feasibility of calcium dobesilate in treatment of renal microvascular injury, the investigators will provide new ideas and theoretical basis for the prevention and treatment of chronic renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Enroll the non dialysis patients with chronic renal failure hospitalized in the Department of Nephrology of the Affiliated Hospital of Xuzhou Medical University.
* According to the glomerular filtration rate, the patients who were not required to be dialysate were at CKD3-5 (GFR between 10 and 59ml/min).

Exclusion Criteria:

* Exclude those patients with diabetes, cardiovascular disease, severe infection, shock, dehydration, abnormal liver function, received glucocorticoid therapy, surgery and emergency dialysis.
* Eliminate those patients with respiratory disease(such as chronic obstructive pulmonary disease, bronchiectasis, asthma), cardiovascular diseases(such as acute and chronic cardiac insufficiency), blood system diseases (such as aplastic anemia, nutritional anemia and polycythemia vera).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
glomerular filtration rate | up to 6 months
  emission computed tomography

SECONDARY OUTCOMES:
serum creatinine | up to 6 months
  intravenous blood sampling
Cystatin C | up to 6 months
  intravenous blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sun, MD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berthet P, Farine JC, Barras JP. Calcium dobesilate: pharmacological profile related to its use in diabetic retinopathy. Int J Clin Pract. 1999 Dec;53(8):631-6. PMID 10692760
- [Background] Tejerina T, Ruiz E. Calcium dobesilate: pharmacology and future approaches. Gen Pharmacol. 1998 Sep;31(3):357-60. doi: 10.1016/s0306-3623(98)00040-8. PMID 9703201
- [Background] Brunet J, Farine JC, Garay RP, Hannaert P. In vitro antioxidant properties of calcium dobesilate. Fundam Clin Pharmacol. 1998;12(2):205-12. doi: 10.1111/j.1472-8206.1998.tb00943.x. PMID 9565776
- [Background] Szabo ME, Haines D, Garay E, Chiavaroli C, Farine JC, Hannaert P, Berta A, Garay RP. Antioxidant properties of calcium dobesilate in ischemic/reperfused diabetic rat retina. Eur J Pharmacol. 2001 Oct 5;428(2):277-86. doi: 10.1016/s0014-2999(01)01196-7. PMID 11675046
- [Background] Brunet J, Farine JC, Garay RP, Hannaert P. Angioprotective action of calcium dobesilate against reactive oxygen species-induced capillary permeability in the rat. Eur J Pharmacol. 1998 Oct 9;358(3):213-20. doi: 10.1016/s0014-2999(98)00604-9. PMID 9822887
- [Background] Padilla E, Ganado P, Sanz M, Zeini M, Ruiz E, Trivino A, Ramirez AI, Salazar JJ, Ramirez JM, Rojas B, Hoz Rd, Tejerina T. Calcium dobesilate attenuates vascular injury and the progression of diabetic retinopathy in streptozotocin-induced diabetic rats. Diabetes Metab Res Rev. 2005 Mar-Apr;21(2):132-42. doi: 10.1002/dmrr.487. PMID 15386814
- [Background] Ruiz E, Lorente R, Tejerina T. Effects of calcium dobesilate on the synthesis of endothelium-dependent relaxing factors in rabbit isolated aorta. Br J Pharmacol. 1997 Jun;121(4):711-6. doi: 10.1038/sj.bjp.0701184. PMID 9208138
- [Background] Lozovskaia EL, Kaplunskii GD, Sapezhinskii II. [Superoxide dismutase activity and photosensitizing properties of 2,5-dihydroxybenzolsulfonate]. Biofizika. 1990 Nov-Dec;35(6):912-6. Russian. PMID 1965686
- [Background] Garay RP, Hannaert P, Chiavaroli C. Calcium dobesilate in the treatment of diabetic retinopathy. Treat Endocrinol. 2005;4(4):221-32. doi: 10.2165/00024677-200504040-00003. PMID 16053339
- [Background] Demirtas S, Caliskan A, Guclu O, Yazici S, Karahan O, Yavuz C, Mavitas B. Can calcium dobesilate be used safely for peripheral microvasculopathies that require neoangiogenesis? Med Sci Monit Basic Res. 2013 Sep 27;19:253-7. doi: 10.12659/MSMBR.889427. PMID 24072135
- [Background] Larsen HW, Sander E, Hoppe R. The value of calcium dobesilate in the treatment of diabetic retinopathy. A controlled clinical trial. Diabetologia. 1977 Apr;13(2):105-9. doi: 10.1007/BF00745136. PMID 323093
- [Background] Allain H, Ramelet AA, Polard E, Bentue-Ferrer D. Safety of calcium dobesilate in chronic venous disease, diabetic retinopathy and haemorrhoids. Drug Saf. 2004;27(9):649-60. doi: 10.2165/00002018-200427090-00003. PMID 15230646
- [Background] Angulo J, Peiro C, Romacho T, Fernandez A, Cuevas B, Gonzalez-Corrochano R, Gimenez-Gallego G, de Tejada IS, Sanchez-Ferrer CF, Cuevas P. Inhibition of vascular endothelial growth factor (VEGF)-induced endothelial proliferation, arterial relaxation, vascular permeability and angiogenesis by dobesilate. Eur J Pharmacol. 2011 Sep 30;667(1-3):153-9. doi: 10.1016/j.ejphar.2011.06.015. Epub 2011 Jun 22. PMID 21703259
- [Background] Barr CC. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive insulin therapy, by The Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. N. Engl. J. Med 342:381-9, 2000. Surv Ophthalmol. 2001 Mar-Apr;45(5):459-60. doi: 10.1016/s0039-6257(01)00187-4. No abstract available. PMID 11274700
- [Background] Ribeiro ML, Seres AI, Carneiro AM, Stur M, Zourdani A, Caillon P, Cunha-Vaz JG; DX-Retinopathy Study Group. Effect of calcium dobesilate on progression of early diabetic retinopathy: a randomised double-blind study. Graefes Arch Clin Exp Ophthalmol. 2006 Dec;244(12):1591-600. doi: 10.1007/s00417-006-0318-2. PMID 16763797
- [Background] Leal EC, Martins J, Voabil P, Liberal J, Chiavaroli C, Bauer J, Cunha-Vaz J, Ambrosio AF. Calcium dobesilate inhibits the alterations in tight junction proteins and leukocyte adhesion to retinal endothelial cells induced by diabetes. Diabetes. 2010 Oct;59(10):2637-45. doi: 10.2337/db09-1421. Epub 2010 Jul 13. PMID 20627932
- [Background] Velpandian T, Nirmal J, Gupta P, Vijayakumar AR, Ghose S. Evaluation of calcium dobesilate for its anti-cataract potential in experimental animal models. Methods Find Exp Clin Pharmacol. 2010 Apr;32(3):171-9. doi: 10.1358/mf.2010.32.3.1423888. PMID 20448859